CLINICAL TRIAL: NCT04354753
Title: AiM COVID for Covid 19 Tracking and Prediction
Status: Completed | Type: Observational
Sponsor: Aarogyam UK (Other)
Collaborators: University of Warwick (Other); Igor Sikorsky Kyiv Polytechnic Institute (Unknown); ClickMedix LLC (Unknown)
Responsible Party: Sponsor
Other Study IDs: AU12
Record Dates: First submitted 2020-04-17; First posted 2020-04-21 (Actual); Last update posted 2020-04-21 (Actual); Status verified 2020-04

CONDITIONS: COVID 19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: No Intervention — No intervention

SUMMARY:
University of Warwick (Coventry, UK) and NTUU "Igor Sikorsky" Kyiv Polytechnic Institute (Kyiv, Ukraine), together with ClickMedix LLC, have developed an app and a chatbot "AiM COVID" for efficient monitoring and mitigation of COVID-19. These products are available for free download on computers and mobile phones. These can be used by a wide range of users from various sectors - patients and people living with them, doctors, nurses, specialists, community health workers, hospitals, clinics, hospital IT staff, MHFA, and insurance companies.

ELIGIBILITY:
Inclusion Criteria:

* Participants 18 and above
* living in UK
* reported with or without symptoms from February 28 to March 28 with community support groups

Exclusion Criteria:

* below 18 years old

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Participants who registered or used any community support services in Leicester
Sampling Method: Non-Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2020-03-28 (Actual); Primary Completion 2020-04-14 (Actual); Study Completion 2020-04-17 (Actual)

PRIMARY OUTCOMES:
Physical symptoms | 1day
  Self reported physical symptoms
Contact History | 14 days
  Contact with suspected, confirmed or ill person
Travel History | 14 days
  Travel to or from overseas

SECONDARY OUTCOMES:
Fever | 1 day
  Self reported body temperature
Headache | 1 day
  Self reported headache using yes/no
Soar Throat | 1 day
  Self reported soar throat using yes/no
Runny nose | 1 day
  Self reported runny nose using yes/no
Cough | 1 day
  Self reported cough using yes/no
Shortness of breath | 1 day
  Self reported shortness of breath symptoms using yes/no
Nausea | 1 day
  Self reported nausea using yes/no
Vomiting | 1 day
  Self reported vomiting using yes/no
Muscle pain | 1 day
  Self reported muscle pain using yes/no
Joint pain | 1 day
  Self reported joint pain using yes/no
Diarrhoea | 1 day
  Self reported Diarrhoea using yes/no
Other | 1 day
  Self reported other symptoms using yes/no
Hospitalisation history | 1 day
  Self reported hospitalisation using yes/no
Co-morbid conditions | 1 day
  Self reported co-morbid conditions using checked box

CONTACTS AND LOCATIONS:
Overall Officials: Vishwesh Kulkarni, Principal Investigator — University of Warwick
Locations (1):
- Aarogyam (UK), Leicester, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided